CLINICAL TRIAL: NCT06119776
Title: Most Total Pancreatectomies for Ductal Adenocarcinoma Can Be Replaced by Whipple Over the Splenic Artery: A Before and After Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202004002RINA
Record Dates: First submitted 2023-08-22; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-08

CONDITIONS: Ductal Adenocarcinoma of the Pancreas
Keywords: Ductal Adenocarcinoma; Pancreatectomies; Whipple

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Patients who underwent Whipple over the splenic artery (WOTSA) as a treatment for PDAC
  Interventions: Procedure: Whipple over the splenic artery
- Control: Patients who underwent total pancreatectomy (TP) as a treatment for PDAC
  Interventions: Procedure: Total pancreatectomy

INTERVENTIONS:
Procedure: Whipple over the splenic artery — Treatment for pancreatic ductal cell adenocarcinoma
  Groups: Study
Procedure: Total pancreatectomy — Treatment for pancreatic ductal cell adenocarcinoma
  Groups: Control

SUMMARY:
Recently, more and more total pancreatectomy (TP) has been performed for pancreatic ductal cell adenocarcinoma (PDCA) which abuts or involves both gastroduodenal and splenic arteries. Warshaw's procedure (spleen-preserving distal pancreatectomy with excision of splenic vessels) has been safely performed for years. Likewise, both pancreatic tail and spleen can be preserved after excision of splenic vessels for leftward extension of pancreatic parenchyma transaction line during Whipple (WOTSA). In that case, TP can be replaced by WOTSA. This uncontrolled before and after study assesses the safety and efficacy of a new technique "Whipple over the splenic artery (WOTSA)" as a treatment for PDAC which traditionally requires total pancreatectomy (TP).

DETAILED DESCRIPTION:
Recently, more and more total pancreatectomy (TP) has been performed for pancreatic ductal cell adenocarcinoma (PDCA) which abuts or involves both gastroduodenal and splenic arteries. Warshaw's procedure (spleen-preserving distal pancreatectomy with excision of splenic vessels) has been safely performed for years. Likewise, both pancreatic tail and spleen can be preserved after excision of splenic vessels for leftward extension of pancreatic parenchyma transaction line during Whipple (WOTSA). In that case, TP can be replaced by WOTSA. This uncontrolled before and after study assesses the safety and efficacy of a new technique "Whipple over the splenic artery (WOTSA)" as a treatment for PDAC which traditionally requires total pancreatectomy (TP).

Methods: The study group comprised 40 consecutive patients who underwent WOTSA for PDAC. Their clinicopathological characteristics and survival were compared with those of a historical control group comprising 30 consecutive patients who underwent TP between.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic ductal cell adenocarcinoma (PDCA) patients

Exclusion Criteria:

* Patient undergoing palliative pancreatectomy, other malignancies with distant metastases
* Vulnerable groups

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pancreatic ductal cell adenocarcinoma (PDCA) patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Clinicopathological characteristics | before
  Measurement of the remnant pancreatic volume
Clinicopathological characteristics | 1 week after the operation
  Measurement of the remnant pancreatic volume

SECONDARY OUTCOMES:
Postoperative chemotherapy and follow-up | 1 month after the operation
  Measurement of the remnant pancreatic volume and physiological parameters

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 day before the operation
  Measurement of the physiological parameters
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months after the operation
  Measurement of the physiological parameters
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months after the operation
  Measurement of the physiological parameters

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided